CLINICAL TRIAL: NCT05788926
Title: A Phase I Dose-escalation Trial of TG6050 Administered by Intravenous Infusion in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Clinical Trial of TG6050 in Patients With Metastatic Non-Small Cell Lung Cancer (Delivir)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not related to safety
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG6050.01
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation of TG6050 (Experimental): Dose escalation with single or repeated administrations of TG6050 by intravenous route in patients with advanced NSCLC.
  Interventions: Drug: TG6050

INTERVENTIONS:
Drug: TG6050 — Oncolytic Vaccinia virus containing genes encoding the human interleukin 12 (IL-12) and an anti-CTLA4 antibody administered at different dose.

SUMMARY:
This is a phase I, open-label, dose-escalation trial of TG6050 administered by single or repeated IV infusion(s).

DETAILED DESCRIPTION:
This clinical trial aims at determining the dose and schedule of administration of TG6050 for further development, primarly based on the assessment of the safety and tolerability of single and repeated IV infusions at escalating doses in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent in accordance with International Conference on Harmonization-Good Clinical Practice and national/local regulations
2. Male or female patient aged 18 to 75 years
3. Histologically confirmed metastatic (stage IV) NSCLC
4. No known oncogenic driver alteration with available targeted therapy, including EGFR, HER2, KRASG12C, MET or BRAFV600E gene mutations and ALK, ROS1, or RET gene fusion/rearrangements. Patients with KRASG12C mutation having received a targeted therapy will be eligible
5. Have received all standard therapeutic options available, including at least 4 months of treatment with an anti-PD1 or PD-L1 monoclonal antibody and doublet platinum-containing chemotherapy
6. Have documented progression not earlier than 4 months after initiation of the anti-PD(L)1 therapy
7. Have at least one measurable lesion according to RECIST 1.1 and at least one lesion amenable to biopsy
8. Expected life expectancy of at least 3 months
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
10. Time from prior immunotherapy or antibody-based therapy to first TG6050 administration of at least 4 weeks, from prior chemotherapy of at least 3 weeks, and from palliative radiotherapy of at least 2 weeks
11. Adequate hematological, hepatic, and renal functions
12. Clearance for trial participation after cardiology consultation and cardiologic investigations
13. Negative pregnancy test in women of childbearing potential (WOCBP)
14. Commitment to use a highly effective contraception method (i.e., with a failure rate of ≤1 % per year) combined with a barrier method (e.g., condom) during TG6050 administration period and at least 3 months after TG6050 administration, in men and WOCBP

Exclusion Criteria:

1. Major surgery within 4 weeks of first TG6050 administration
2. Prior treatment with ipilimumab
3. Prior treatment with an oncolytic virus
4. Prior treatment with another investigational agent within 4 weeks of first TG6050 administration
5. Immunodeficiency due to underlying illness and/or immune-suppressive medication
6. Uncontrolled intercurrent illness
7. Active auto-immune disease except hypothyroidism or type I diabetes only requiring hormone replacement therapy
8. Brain metastases, unless treated and stable for at least 4 weeks after medical imaging assessment
9. Other malignancies than NSCLC except cutaneous basal cell carcinoma and in situ carcinoma of the uterine cervix, unless complete remission for at least 5 years prior to trial entry and no therapy required during the trial
10. Ongoing antiviral therapy active on vaccinia virus (VV), e.g., ribavirin, interferon/pegylated interferon
11. History of monkeypox infection or anti-monkeypox vaccination
12. History of severe exfoliative skin conditions
13. History of grade ≥ 3 auto-immune manifestations related to ICI therapy
14. History of severe systemic reaction or side-effect after a smallpox vaccination
15. History of solid organ or allogeneic stem cell transplantation
16. Known hypersensitivity to eggs or any TG6050 excipients
17. Positive test for hepatitis C virus (HCV) or hepatitis B virus (HBV) indicating acute or chronic infection
18. Live virus vaccination within 28 days of TG6050 administration
19. COVID-19 vaccination or infection within 14 days of TG6050 administration
20. Breastfeeding woman
21. Any medical, familial, sociological, or psychiatric condition that in the opinion of the investigator would prohibit inclusion in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Adverse Event reported per NCI-CTCAE v5.0) | Up to 5 years
  Incidence of Adverse Event reported per NCI-CTCAE v5.0, Dose limiting toxicity, Maximal tolerated dose, Maximum feasible dose and Serious Adverse Events.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 1 year
  Proportion of patients whose best response during their participation in the trial is either complete response (CR) or partial response (PR)
4-month disease control rate | Up to 4 months
  Proportion of patients whose tumor assessment at 4 months is either complete response (CR), partial response (PR), or stable disease (SD)
Overall disease control rate (DCR) | Up to 1 year
  Proportion of patients whose tumor assessment is either complete response (CR), partial response (PR), or stable disease (SD) during their trial participation
Progression-free survival (PFS) | Up to 1 year
  Time from the first TG6050 infusion to documented tumor progression or death due to any cause.
Overall survival (OS) | Up to 1 year
  Time from the first TG6050 infusion to death due to any cause.
Duration of overall response (DoR) | Up to 1 year
  Time from the first documented response (complete response (CR) or partial response (PR)) to documented tumor progression or death due to underlying cancer.
Molecular responses (MR) | Up to 1 year
  Circulating tumor DNA (ctDNA) levels and changes over time

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - Hôpital Timone, Marseille
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azar F, Deforges J, Demeusoit C, Kleinpeter P, Remy C, Silvestre N, Foloppe J, Fend L, Spring-Giusti C, Quemeneur E, Marchand JB. TG6050, an oncolytic vaccinia virus encoding interleukin-12 and anti-CTLA-4 antibody, favors tumor regression via profound immune remodeling of the tumor microenvironment. J Immunother Cancer. 2024 Jul 25;12(7):e009302. doi: 10.1136/jitc-2024-009302. PMID 39060022